CLINICAL TRIAL: NCT01432392
Title: A Prospective, Observational Study to Describe Symptom Control and Impact on Daily Life in Patients With Gastroesophageal Reflux Disease (GERD)
Brief Title: Symptom Control and Impact on Daily Life in Patients With Gastroesophageal Reflux Disease
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-GBG-XXX-2011/1
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: gastroesophageal reflux disease; GERD questionnaire; primary care setting
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
The purpose of this study is to evaluate the impact of gastroesophageal reflux disease (GERD) treatment in primary care setting on symptom control and daily life in symptomatic GERD patients, using both GERD questionnaire and clinical symptoms assessment

DETAILED DESCRIPTION:
A prospective, observational study to describe symptom control and impact on daily life in patients with gastroesophageal reflux disease (GERD)

ELIGIBILITY:
Inclusion Criteria:

* Patients known or newly diagnosed with GERD
* Patients with typical GERD symptoms as heartburn and regurgitation for ≥2 days in the previous week
* Patients, currently not treated with a proton pump inhibitor

Exclusion Criteria:

* Patients who have been receiving treatment with non-steroidal antiinflammatory drugs within two weeks prior the inclusion in the study
* Patients with medical history of surgery of the esophagus, stomach or duodenum
* Pregnant or nursing females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care setting
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Percent change in intensity and frequency for each of typical GERD symptoms from baseline to week 4-6 | Day 0 to week 4-6
Changes in GERD questionnaire(GERD-Q) scores from baseline to week 4-6 | Day 0 to week 4-6

SECONDARY OUTCOMES:
To evaluate the correlation between GERD-Q scores and symptom scores | two times

CONTACTS AND LOCATIONS:
Locations (2):
- Bulgaria (2):
  - Sofia
  - Varna